CLINICAL TRIAL: NCT00896558
Title: A Double-Blind, Parallel, Randomized, Placebo-Controlled, Repeat Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK1322322 in Healthy Subjects
Brief Title: A Repeat Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK1322322 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 112668
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Infections, Bacterial
Keywords: GSK1322322, repeat dose, healthy subjects, elderly, drug-drug interaction, probe, midazolam, double-blind
MeSH Terms: conditions — Bacterial Infections | interventions — GSK1322322; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort A (Experimental): A single AM dose of GSK1322322/placebo on Day 1, no dosing on Day 2, and BID dosing on Days 3-12.
  Interventions: Drug: GSK1322322/placebo
- Cohort B (Experimental): Subjects will receive a single AM dose of GSK1322322/placebo on Day 1, no dosing on Day 2, and BID dosing on Days 3-12.
  Interventions: Drug: GSK1322322/placebo
- Cohort C (Experimental): Subjects in the probe cohort will receive a single AM dose of GSK1322322/placebo on Day 1, no dosing on Day 2, and BID dosing on Days 3-12. All subjects will receive a single dose of midazolam alone on Day -1, and co-administered with the morning dose of GSK1322322/placebo on Day 1 and Day 12.
  Interventions: Drug: GSK1322322/placebo; Drug: GSK1322322/placebo and midazolam
- Cohort D (Experimental): Subjects will receive a single AM dose of GSK1322322/placebo on Day 1, no dosing on Day 2, and BID dosing on Days 3-12.
  Interventions: Drug: GSK1322322/placebo
- Cohort E (Experimental): Subjects will receive a single AM dose of GSK1322322/placebo on Day 1, no dosing on Day 2, and BID dosing on Days 3-12.
  Interventions: Drug: GSK1322322/placebo

INTERVENTIONS:
Drug: GSK1322322/placebo — GSK1322322/placebo escalating doses from 500mg to 1500mg
Drug: GSK1322322/placebo and midazolam — GSK1322322/placebo and 5mg midazolam
  Arms: Cohort C

SUMMARY:
This study will be the first repeat dose administration of GSK1322322 to investigate safety, tolerability, and pharmacokinetics in healthy subjects as well as elderly volunteer subjects. The study will also include a P450 probe drug (midazolam) to evaluate the effect of GSK1322322 to inhibit or induce CYP3A4 substrates.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent (except for elderly cohort-Part B, see #8 below)..
* A female is eligible to enter and participate in this study if she is of non-childbearing potential
* Male subjects must agree to use one of the contraception methods in the protocol
* Body weight greater than or equal to 50 kg and body mass index between 18.5-29.9 kg/m2 inclusive
* Capable of giving written informed consent
* QTcB less than 450 msec; or QTc less than 480 msec in subjects with Bundle Branch Block on Screening ECG
* Part B/Cohort E Elderly cohort: The subject is greater than 65 years of age.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined in the protocol
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive human chorionic gonadotropin test at screening or prior to dosing.
* Lactating females.
* Subjects who have asthma or a history of asthma within the past 6 months.
* History of smoking or history of regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, satsuma, ugli, tangerine, and tangelo, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* For probe cohort in Part A: any condition or symptom contraindicated for administration of midazolam including acute narrow-angle or open-angle glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-05-11 (Actual); Primary Completion 2009-09-25 (Actual); Study Completion 2009-09-25 (Actual)

PRIMARY OUTCOMES:
GSK1322322 safety parameters, adverse events , absolute values and changes over time of clinical lab testing, vital signs, electrocardiogram | 6 weeks
GSK1322322 pharmacokinetic parameters following single dose administration on Day 1 and following repeat administration where applicable on Day 7 and Day 12. | 15 days

SECONDARY OUTCOMES:
PK for midazolam with and without GSK1322322 | 15 days
Blood PK for GSK1322322 | 15 days
Urine PK for GSK1322322 | 15 days
GSK1322322 Age Effect on PK Blood and Urine | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Naderer OJ, Dumont E, Zhu J, Kurtinecz M, Jones LS. Safety, tolerability and pharmacokinetics of repeat dosing of the antibiotic GSK1322322, a peptide deformylase inhibitor: a randomized placebo-controlled study. J Antimicrob Chemother. 2013 Aug;68(8):1901-9. doi: 10.1093/jac/dkt097. Epub 2013 Apr 3. PMID 23557930
- See also: Results for study 112668 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112668?search=study&study_ids=112668#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112668 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112668 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112668 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112668 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112668 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112668 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112668 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register